CLINICAL TRIAL: NCT01131026
Title: A Monocentric, Open-label, Efficacy and Safety Evaluation Study of the Triple Therapy of 500 mg Levofloxacin, 1000 mg Amoxicillin and 30 mg Lansoprazole on Helicobacter Pylori Eradication in 60 Patients Infected With H. Pylori
Brief Title: Efficacy and Safety Evaluation of Levofloxacin Triple Therapy for Helicobacter Pylori Eradication
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Deva Holding A.S. (Industry)
Collaborators: TNC Ilac Arastirma Gelistirme Danismanlik San. ve Tic. Ltd. Sti. (Other); TC Erciyes University (Other)
Responsible Party: Prof. Dr. R. Serdar Alpan, MD, PhD, MSc, TNC İlac Arastirma Gelistirme Danismanlik San. ve Tic. Ltd. Sti.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DV-09-0015
Record Dates: First submitted 2010-05-12; First posted 2010-05-26 (Estimated); Last update posted 2011-08-09 (Estimated); Status verified 2011-08

CONDITIONS: Helicobacter Pylori Infection
Keywords: Helicobacter pylori; levofloxacin; amoxicillin; lansoprazole; efficacy; safety; triple therapy
MeSH Terms: interventions — Levofloxacin; Tablets; Amoxicillin; Lansoprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Levofloxacin — tablet, 500 mg, once a day for ten days
  Other Names: Floxilevo 500 mg Tablet
Drug: Amoxicillin — tablet, 1000 mg, once a day for ten days
  Other Names: Dentamax 1 gr Tablet
Drug: Lansoprazole — capsule, 30 mg, twice a day for ten days
  Other Names: Degastrol 30 mg Capsule

SUMMARY:
Today, although the triple treatment with clarithromycin accepted as the primary treatment for Helicobacter pylori infection eradication is well tolerated, the eradication has been decreased to 65 %. However, the eradication resulting from TRIOL treatment with levofloxacin is expected to be 75 % or higher. If the target results can be reached, it will be concluded that TRIOL treatment with levofloxacin will be an alternative to the triple treatment with clarithromycin as the primary treatment.

DETAILED DESCRIPTION:
The primary end point in this study is appointed to be "Helicobacter pylori infection eradication with TRIOL treatment" and the secondary end point as "safety". The study involves the investigation of the efficacy and safety of the triple treatment consisting of 500 mg levofloxacin, 1000 mg amoxicillin and 30 mg lansoprazole on Helicobacter pylori eradication in 60 patients with Helicobacter pylori infection.

ELIGIBILITY:
Inclusion Criteria:

* Consenting to an endoscopy
* Signing the informed consent form
* Not receiving Helicobacter pylori eradication treatment before
* Showing Helicobacter pylori infection by rapid urease test and/or Giemsa staining
* Being older than 18 years of age

Exclusion Criteria:

* Being younger than 18 years of age
* Receiving H. pylori eradication treatment previously
* Having gastrectomy or vagotomy in medical history
* Having gastric malignancy, including adenocarcinoma and lymphoma
* Having other severe malignant disease
* Previously having allergic reaction to antibiotics (amoxicillin, levofloxacin) and proton pump inhibitors (lansoprazole)
* Using prompt pump inhibitors (lansoprazole) and antibiotics (amoxicillin, clarithromycin, levofloxacin) in the last 4 weeks
* Having active upper GI bleeding in the last week
* Being pregnant or lactating
* Taking long term high dosages of aspirin, corticosteroid and other NSAIDs in the last 4 weeks
* Taking any antibiotics or proton pump inhibitors other than the study medication during the study period
* Taking antacids and/or H2-blockers during the study period
* Taking bismuth compounds within four weeks prior to and during the study period
* Having dysphasia or vomiting as major symptoms
* Having psychiatric, neurological, or behavioral disorders that may interfere with the conduct or interpretation of the study
* Having severe concomitant disease of the cardiovascular, pulmonic, hepatic, renal, hematological, lymphatic, metabolic, and endocrine system.
* Having known uncontrolled hypertension
* Being immunocompromised
* Showing clinically significant abnormal vital signs
* Having clinically significant abnormal ECG findings
* Presenting clinically significant abnormal laboratory data at screening, or any abnormal laboratory value that could interfere with the assessment of safety
* Being exposed to any investigational drug within 30 days prior to screening
* Having known hypersensitivity to or contraindication against fluoroquinolones.
* Having current diagnosis or known history of substance abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2010-06; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Helicobacter pylori infection eradication | 6 weeks
  After 6 weeks from the end of the TRIOL treatment, demonstrating the ratio of patients who do not develop Helicobacter pylori infection by rapid urease test and Giemsa staining.

SECONDARY OUTCOMES:
Safety | 6 weeks
  During the study all patients will be examined at the determined timepoints in the protocol in regard to any type of clinical adverse event. These examinations involve clinical and laboratory examinations of which the results will be recorded in the final study report and discussed with respect to the current literature.

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Yucesoy, MD, Principal Investigator — Kayseri, Erciyes University School of Medicine Hospital, Department of Internal Medicine and Gastroenterology; Recep S Alpan, MD, PhD, MSc, Study Director — TNC Pharmaceuticals Research, Development and Consultancy Ltd.
Locations (1):
- Erciyes University School of Medicine Hospital, Department of Internal Medicine and Gastroenterology, Kayseri, Turkey (Türkiye)